CLINICAL TRIAL: NCT01819350
Title: Avaliação in Vivo do Potencial cariogênico e Erosivo de Bebidas e Medicamentos pediátricos líquidos Intra-orais
Brief Title: In Vivo Study of Sucrose and Liquid Oral Pediatric Medicines of Long-term Effect on Dental Biofilm pH
Acronym: SPMedicines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Fabio Correia Sampaio, PhD, Federal University of Paraíba
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: SOPM-UFPB
Record Dates: First submitted 2013-03-24; First posted 2013-03-27 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Dental Biofilm pH
Keywords: Dental caries; Sucrose; Oral administration; Ion Concentration of Hydrogen; Pediatric medicines
MeSH Terms: conditions — Dental Caries | interventions — HLA-G Antigens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- G4 and G5 (Experimental): Application of antibiotic group of pediatric medicines and control group (sucrose 10 %)on dental biofilm.
  Interventions: Other: G4 and G5
- G1, G2 and G3 (Experimental): Application of Nutritional, Respiratory and Endocrine groups medicines pediatric on dental biofilm
  Interventions: Other: G1, G2 and G3

INTERVENTIONS:
Other: G1, G2 and G3 — Nutritional, respiratory and endocrine group applicated 12 subjects
  Arms: G1, G2 and G3
Other: G4 and G5 — Application of trhree pediadic medidines of antibiotic group on dental biofilm 12 subjects
  Arms: G4 and G5

SUMMARY:
The aims of this study were to determine the sucrose and liquid oral pediatric medicines of long-term effect on dental biofilm pH to evaluate the cariogenic potential in vivo.

DETAILED DESCRIPTION:
Te study was carried out with 12 subjects that were refrained from brushing their teeth for 28 h and did not eat or drink for at least 3 h prior to each appointment. Dental biofilm pH was measured in the cervical and proximal regions of anterior teeth with beetrode-type microelectrode coupled to a potentiometer. The biofilm was submitted nine paediatric medicines a long term and sucrose (negative control). pH measurements were taken at baseline to determine resting plaque pH and at time interval 5, 10, 15, 20, 25 and 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 22 years;
* Having Oral hygiene adequate (OHI<1.1);
* Having 20 natural teeth incluing molar;
* Not havind oral disease.

Exclusion Criteria:

* Biofilm baseline pH > 5,5;
* Not signature consent term;
* Using orthodontic appliance;
* Having used medicines last 3 months;
* Pregant woman.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of group respiratory, nutritional and endocrine pediatric medicines effect on dental biofilm pH | 6 months
  pH was measured in the cervical and proximal regions of anterior teeth dental biofilm with beetrode-type microelectrode coupled to a potentiometer

SECONDARY OUTCOMES:
Evaluation of sucrose antibiotic group and control negative group effect on dental biofilm | 12 months
  The biofilm was submitted antibiotic group and negative control group. pH measurements were taken at baseline to determine resting plaque pH and at time interval 5, 10, 15, 20, 25 and 30 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Paraíba, João Pessoa, Paraíba, Brazil